CLINICAL TRIAL: NCT05379387
Title: Health-related Quality of Life and Late Effects Among SURVivors of Cancer in Adolescence and Young Adulthood: The SURVAYA Study
Status: Completed | Type: Observational
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: IRBd18122
Record Dates: First submitted 2022-05-13; First posted 2022-05-18 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Quality of Life; Late Effect; Survivorship; Lifestyle; Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Rationale: Adolescent and young adult (AYA) cancer survivors, diagnosed between 18-39 years, much more than children, suffer from delay in diagnosis, lack of centralization of care, age-adjusted expertise and follow-up care. The distribution of tumor types, biology, risk factors, developmental challenges and treatment regimens are different in AYAs compared to children. Therefore findings derived from childhood cancer survivors cannot be extrapolated to AYAs. Likewise, several large tumor-specific cohort studies exist that do not specifically address unique AYA age-specific issues. Globally, so far, the identification of AYA patient subgroups that might be more susceptible to poor health outcomes has not been systematically addressed. The role of sociodemographic and treatment-associated risks, external exposures (e.g. lifestyle) and host factors (e.g. genetic); or combinations of influences for impaired (age-specific) health outcomes, remains largely unknown. Understanding who is at risk and why, will support the development of evidence-based AYA prevention, treatment and supportive care programs and guidelines.

Objective: To examine the prevalence, risk factors and mechanisms of impaired health outcomes (health-related quality of life and late effects) among a population-based sample of AYA cancer survivors. Study design: Retrospective, population-based, observational cohort study.

Study population: AYA cancer survivors, diagnosed at age 18-39 years between 1999-2015, identified from the Netherlands Cancer Registry (NCR), and alive 5-20 year after diagnosis Main study parameters/endpoints: Health-related quality of life; late effects

ELIGIBILITY:
Inclusion Criteria:

* Pathological confirmed cancer diagnosis;
* Age 18 - 39 years at time of first cancer diagnosis;
* Provide written informed consent.
* Treated in an Academic hospital or Netherlands Cancer Institute

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All AYA cancer patients, diagnosed at age 18-39 years and treated in one of the participating hospitals
Sampling Method: Probability Sample
Enrollment: 4000 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Health related quality of life | Day 1
  The EORTC QLQ-C30 is a 30-item HRQoL questionnaire consisting of five functional scales (physical, role, cognitive, emotional and social), a global quality of life scales, symptom scales (fatigue, pain, nausea and vomiting) and a number of single items assessing common symptoms (dyspnea, loss of appetite, sleep disturbance, constipation and diarrhea) and perceived financial impact of the disease. After linear transformation, all scales and single item measures range in score from 0-100. A higher score on the functional scales and global QoL means better functioning and HRQoL, whereas a higher score on the symptom scales means more complaints.

CONTACTS AND LOCATIONS:
Overall Officials: Winette van der Graaf, Prof, Study Director — Netherlands Cancer Institute - Antoni van Leeuwenhoek Hospital (NKI-AvL)
Locations (1):
- Antoni van Leeuwenhoekziekenhuis, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Janssen SHM, Vlooswijk C, Bijlsma RM, Kaal SEJ, Kerst JM, Tromp JM, Bos MEMM, van der Hulle T, Lalisang RI, Nuver J, Kouwenhoven MCM, van der Graaf WTA, Husson O. Health-related quality of life of long-term adolescent and young adult (AYA) cancer survivors compared to a matched normative population: results of the SURVAYA study. J Cancer Surviv. 2025 Jun 17. doi: 10.1007/s11764-025-01818-0. Online ahead of print. PMID 40528140
- [Derived] Janssen SHM, Vlooswijk C, Bijlsma RM, Kaal SEJ, Kerst JM, Tromp JM, Bos MEMM, van der Hulle T, Lalisang RI, Nuver J, Kouwenhoven MCM, van der Graaf WTA, Husson O. Health-related conditions among long-term cancer survivors diagnosed in adolescence and young adulthood (AYA): results of the SURVAYA study. J Cancer Surviv. 2025 Dec;19(6):1821-1834. doi: 10.1007/s11764-024-01597-0. Epub 2024 May 13. PMID 38740702